CLINICAL TRIAL: NCT00366496
Title: Comparison of Visual Outcomes, Wavefront Analysis, Contrast Sensitivity and Glare Testing Following Cataract Extraction Between Acrysof Single-Piece IOL and Acrysof WF
Brief Title: Surgical Outcomes After Routine Cataract Extraction & Implantation of a Conventional or Spheric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-05-004
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2005-07

CONDITIONS: Cataract Extraction

INTERVENTIONS:
Device: Acrysof single piece (SA60AT)
Device: Acrysof IQ (SN60WF)

SUMMARY:
To determine quality of vision post cataract extraction and intraocular lens (IOL) implantation of 2 different acrylic intraocular lenses: Acrysof® Single-Piece IOL and Acrysof® WF, through evaluation of contrast sensitivity, glare testing, visual outcomes, wavefront, corneal topography, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral cataract
* Eligible for phacoemulsification with primary implantation of a posterior chamber IOL. If bilateral, patient will receive the same IOL than the fellow eye.
* Expected maximum of 4 weeks and minimum of 1 week interval between primary and second eye surgeries when bilateral.
* Best corrected visual acuity (BCVA) should be no better than 20/40 in the presence of a glare source using Snellen visual acuity. In the Snellen visual acuity chart, better than 20/40 will be at least 3 letters read correctly in the 20/30 line.
* Naturally dilated pupil (in dim light) ≥ 4.0 mm in both eyes.

Exclusion Criteria:

* Preoperative ocular pathology potentially affecting visual acuity
* Previous intraocular or corneal surgery.
* Keratometric astigmatism exceeding 1.5 diopters.
* Planned postoperative refraction for mono-vision.
* Current contact lens usage.
* Other ocular surgery at the time of the cataract extraction.
* Uncontrolled diabetes.
* Any neurological condition that might interfere with performance of required test.
* Auto-immune deficiency disease.
* Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Use of any systemic or topical drug known to interfere with visual performance.

Surgical Exclusion Criteria

* Significant anterior chamber bleeding.
* Detached Descemet's membrane
* Iris damage
* Posterior capsule rupture
* Radial tear in capsulorhexis
* Vitreous loss
* Zonular rupture.
* Use of corneal sutures for more than 1 week.

Post-implantation Exclusion Criteria

* Haptic not in the capsular bag.
* Descentration of the IOL of more than 1.0 mm
* Ocular pathologies potentially affecting visual acuity that were not evident prior to surgery.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-05

PRIMARY OUTCOMES:
Contrast sensitivity
Visual acuity

SECONDARY OUTCOMES:
Induction of hight order aberrations
Corneal topography
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina